CLINICAL TRIAL: NCT00161369
Title: Contribution of Homocysteine and Asymmetric Dimethylarginine to Atherosclerosis and Cardiovascular Events in Maintenance Hemodialysis Patients
Brief Title: Effect of Homocysteine and Asymmetric Dimethylarginine on Cardiovascular Events in Hemodialysis Patients
Status: Completed | Type: Observational
Sponsor: University of Shizuoka (Other)
Collaborators: Maruyama Memorial General Hospital (Other); Hamamatsu University (Other)
Other Study IDs: CT2005001
Record Dates: First submitted 2005-09-09; First posted 2005-09-12 (Estimated); Last update posted 2005-10-21 (Estimated); Status verified 2005-10

CONDITIONS: Chronic Renal Failure; Hemodialysis; Atherosclerosis
Keywords: homocysteine; asymmetric dimethylarginine; atherosclerosis; cardiovascular event; hemodialysis
MeSH Terms: conditions — Kidney Failure, Chronic; Atherosclerosis

STUDY DESIGN:
Observational Model: Defined Population | Time Perspective: Prospective

SUMMARY:
Homocysteine (Hcy) and asymmetric dimethylarginine (ADMA) have recently been recognized as potential risk factors for atherosclerosis in the general population, and the metabolism of each of these substances seems to be closely related. This study investigates the association between these substances, and whether elevated serum levels of Hcy and ADMA would be related to a high risk of atherosclerosis and cardiovascular events in maintenance hemodialysis (HD) patients.

DETAILED DESCRIPTION:
Objective- Homocysteine (Hcy) and asymmetric dimethylarginine (ADMA) have recently been recognized as potential risk factors for atherosclerosis in the general population, and the metabolism of each of these substances seems to be closely related. This study investigates the association between these substances, and whether elevated serum levels of Hcy and ADMA would be related to a high risk of atherosclerosis and cardiovascular events in maintenance hemodialysis (HD) patients.

Methods- The subjects were recruited from both day-time and night-time HD patients at Maruyama Hospital. The study inclusion criteria were those patients who had been receiving hemodialysis therapy for more than 6 months, were in a stable condition and were under 70 years old. The degree of atherosclerosis was evaluated by four indices involving the carotid artery intima-media thickness (IMT), carotid artery plaque, percentile of calcification index in the abdominal aortic wall (ACI) and elongation of the thoracic aorta. At the same time, plasma Hcy and ADMA were measured. After the initial laboratory examination and evaluation of the degree of atherosclerosis, all the patients were followed up for 5 years.

ELIGIBILITY:
Inclusion Criteria:

* The study inclusion criteria were those patients who had been receiving hemodialysis therapy for more than 6 months, were in a stable condition and were under 70 years old.

Exclusion Criteria:

* Any patients showing signs of heart failure or a history of such apparent cardiovascular diseases as myocardial infarction, cardiac valve diseases and stroke were excluded.

Max Age: 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 200
Dates: Start 2000-04; Study Completion 2005-03

CONTACTS AND LOCATIONS:
Overall Officials: Hiromichi Kumagai, MD, Study Chair — University of Shizuoka
Locations (1):
- University of Shizuoka, Shizuoka, Shizuoka, Japan